CLINICAL TRIAL: NCT00420251
Title: Recombinant Human Growth Hormone Treatment in Juvenile Idiopathic Arthritis: Controlled Study on the Effect on Growth and Bone Development
Brief Title: Efficacy and Safety of Growth Hormone Treatment in Juvenile Idiopathic Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13042004
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2007-01-11 (Estimated); Status verified 2007-01

CONDITIONS: Juvenile Idiopathic Arthritis; Still Disease, Juvenile-Onset
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Human Growth Hormone

INTERVENTIONS:
Drug: Genotropin

SUMMARY:
Growth retardation is well known in patients with severe forms of juvenile idiopathic arthritis. Especially those who were under additional treatment with glucocorticoids for high disease activity. The hypothesis is, that treatment with growth hormone can, at leat in part, overcome growth hormone resistance state and increase final height. In a controlled study we follow patients with juvenile idiopathic arthritis with and without growth hormone treatment until final height. Additionally, we are interested in bone density development in those treated with growth hormone.

DETAILED DESCRIPTION:
Growth retardation is well known in patients with severe forms of juvenile idiopathic arthritis. Especially those who were under additional treatment with glucocorticoids for high disease activity. This is the case in patients with a polyarticular and a systemic form of juvenile idiopathic arthritis. The permanent consequence is short stature at final height. Up to 30% of these patients will have a final height below the 3rd percentile, even after discontinuation of glucocorticoid treatment. The hypothesis is, that treatment with growth hormone can, at leat in part, overcome growth hormone resistance state and increase final height. In a controlled study we follow patients with juvenile idiopathic arthritis with and without growth hormone treatment until final height. From safety aspects we were interested in the effect of growth hormone on the disease activity. Additionally, we are interested in bone density development in those treated with growth hormone up to final height.

ELIGIBILITY:
Inclusion Criteria:

* Polyarticular or systemic juvenile idiopathic arthritis,
* Growth velocity below the 25th percentile and or short stature ,
* Treatment with glucocorticoids for at least the previous 6 months before inclusion,
* Prepubertal stage,
* Bone age below 10 in girls and 12 in boys,
* Growth hormone levels after stimulation with clonidine or arginine above 10 ng/ml

Exclusion Criteria:

* Previous treatment with growth hormone,
* Endocrinopathy,
* Additional chronic disease beside juvenile idiopathic arthritis,
* Malignant disase,
* Chromosomal aberration or othe syndromal disease,
* Previous treatment with Oxandrolone,
* Small for gestational age,
* Elevated fasting glucose level

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50
Dates: Start 1996-03; Study Completion 2006-07

PRIMARY OUTCOMES:
Final height

SECONDARY OUTCOMES:
Bone geometry and density

CONTACTS AND LOCATIONS:
Overall Officials: Susanne M Bechtold, MD, Principal Investigator — University Children´s Hospital, Munich
Locations (1):
- Center For Rheumatic Diseases in Childhood, Garmisch-Partenkirchen, Germany

REFERENCES:
- [Result] Bechtold S, Ripperger P, Muhlbayer D, Truckenbrodt H, Hafner R, Butenandt O, Schwarz HP. GH therapy in juvenile chronic arthritis: results of a two-year controlled study on growth and bone. J Clin Endocrinol Metab. 2001 Dec;86(12):5737-44. doi: 10.1210/jcem.86.12.8083. PMID 11739431
- [Result] Bechtold S, Ripperger P, Hafner R, Said E, Schwarz HP. Growth hormone improves height in patients with juvenile idiopathic arthritis: 4-year data of a controlled study. J Pediatr. 2003 Oct;143(4):512-9. doi: 10.1067/S0022-3476(03)00390-1. PMID 14571231